CLINICAL TRIAL: NCT02403726
Title: Osteoporosis Associated Vertebral Fractures - Medical and Socio-economic Aspects in Austria
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, MD, Medical University of Vienna
Other Study IDs: 2011/896
Record Dates: First submitted 2015-03-20; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- osteoporosis associated vertebral fractures: Analyzation of demographic, medical, gender and socio-economic aspects of osteoporosis associated vertebral fractures.
  Interventions: Procedure: Operation; Procedure: Non-operative treatment

INTERVENTIONS:
Procedure: Operation — Analyzation of demographic, medical, gender and socio-economic aspects of osteoporosis associated vertebral fractures treated with operation.
Procedure: Non-operative treatment — Analyzation of demographic, medical, gender and socio-economic aspects of osteoporosis associated vertebral fractures treated with non-operative treatment.

SUMMARY:
The purposes of this study were to analyse demographic, medical, gender and socio-economic aspects of osteoporosis associated vertebral fractures.

ELIGIBILITY:
Inclusion Criteria:

-patients older than 50 years of age with vertebral fractures at the thoracic or lumbar spine caused by a low-energy trauma or without any trauma, or with vertebral fractures at the thoracic or lumbar spine with typical osteoporotic deformity of the vertebrae (wedge, fish, or flat)

Exclusion Criteria:

* patients younger than 50 years of age
* vertebral fractures at the cervical spine
* vertebral fractures at the thoracic or lumbar spine caused by a high-energy trauma (motor-vehicle accident, sports-related accident, fall from a considerable height)
* patients suffering from a malignancy, making a pathological fracture presumably, patients with vertebral fractures, whose dataset of follow-up monitoring was lacking, to make an evaluation of osteoporotic involvement impossible

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was a retrospective case series of 694 patients, in which the fracture was caused due to primary or secondary osteoporosis, and who were treated at the department of trauma surgery at our level-I trauma center.
Sampling Method: Non-Probability Sample
Enrollment: 694 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
demographic aspects | at least two year follow up
  demographic aspects (age, social status) of osteoporosis associated vertebral fractures treated with either operation or non operative treatment
gender aspects | at least two year follow up
  gender aspects (sex) of osteoporosis associated vertebral fractures treated with either operation or non operative treatment
socio economic aspects | at least two year follow up
  socio-economic aspects (cost ratio) of osteoporosis associated vertebral fractures treated with either operation or non operative treatment